CLINICAL TRIAL: NCT02050581
Title: "A Chart Review of Rituximab Plus Repeated Cycles of Dexamethasone for the Treatment of Relapsed/Refractory ITP:"
Brief Title: A Chart Review of Rituximab Plus Repeated Cycles of Dexamethasone
Acronym: Dex/Rituxan
Status: Terminated | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1012011459
Record Dates: First submitted 2014-01-13; First posted 2014-01-31 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Idiopathic Thrombocytopenia Purpura
Keywords: Platelets are a part of the blood hat helps with clotting; ITP idiopathic thrombocytopenia purpura low platelet count
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
In this prospective and retrospective chart review, investigators will evaluate the response rates and duration of response for patients with relapsed and refractory idiopathic thrombocytopenic purpura (ITP) who have been treated with rituximab and repeated courses of dexamethasone. Investigators will also evaluate observed toxicities of the combination, and characteristics associated with response.

DETAILED DESCRIPTION:
Patients with idiopathic thrombocytopenic purpura (ITP) usually respond with an increase in platelet count after treatment with steroids, but most patients will experience recurrence.Rituximab has been a useful treatment for patients with recurrent ITP; many hundreds of patients have been treated. 30-40% of patients will achieve a complete remission (CR: platelet count >150 x 109/l) with initial treatment. However, most patients will relapse between 1 and 3 years from initial treatment suggesting that long-term "cures" only occur in 20% of the initial patients. An increased rate of durable CRs is therefore a desirable goal. One approach would be to use rituximab maintenance; however, this strategy results in long term B cell suppression. Dexamethasone has also been used to achieve "cure" in ITP, especially in adults at or near diagnosis. An initial study suggested that approximately 50% of patients would achieve a long-term response with only one 4-day cycle of high dose (40 mg/day) dexamethasone. A follow up study suggested that 3-4 cycles of dexamethasone would be better than 1 cycle. Finally, a recent publication suggested that rituximab plus one cycle of dexamethasone was superior to dexamethasone alone, with a > 50% CR rate at 6 months. Based on the published activity of rituximab and dexamethasone in this disorder, some patients have received treatment with combined dexamethasone and rituximab. We will review the data of those patients who have received more than one course of dexamethasone together with rituximab for relapsed or refractory ITP in order to determine the response rate, duration of response, toxicity of the combination, and clinical predictors of response in this group.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be diagnosed with ITP.
2. Subjects must be 3 years old or older
3. Subjects must have a platelet count less than 40,000/uL at initiation of treatment regimen or inability to discontinue maintenance treatments such as intravenous immunoglobulin (IVIG), corticosteroids, azathioprine, and/or a thrombopoietin receptor agonist.

Exclusion Criteria:

1. Subjects who have not been diagnosed with ITP. 2 Subjects who are younger than 3 years old 3. Subjects who have a medical condition that would be adversely affected by high dose steroids

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received more than one course of dexamethasone together with rituximab for relapsed or refractory ITP.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2011-01; Primary Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
An increase in Platelet count | 8 weeks
  An increase in Platelet count after 8 weeks on treatment

SECONDARY OUTCOMES:
Achieve a complete or partial response to treatment | Within an average of 12 weeks
  Investigators hope patients will achieve a complete response (a platelet count greater than or equal to 100,000/uL) or a partial response (a platelet count between 50,000/uL and 99,000/uL) not due to rescue medication within an average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James B Bussel, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bussel JB, Lee CS, Seery C, Imahiyerobo AA, Thompson MV, Catellier D, Turenne IG, Patel VL, Basciano PA, Elstrom RL, Ghanima W. Rituximab and three dexamethasone cycles provide responses similar to splenectomy in women and those with immune thrombocytopenia of less than two years duration. Haematologica. 2014 Jul;99(7):1264-71. doi: 10.3324/haematol.2013.103291. Epub 2014 Apr 18. PMID 24747949